CLINICAL TRIAL: NCT02022969
Title: Detection of SpO2-oscillations Caused by Cyclic Recruitment and Derecruitment of Low Ventilated Areas in the Lung (Atelectasis) During Mechanical Ventilation
Brief Title: Detection of SpO2-oscillations of Low Ventilated Areas
Acronym: MAS
Status: Withdrawn | Type: Observational
Why Stopped: Personell
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ass.-Prof. PD Dr. Klaus Ulrich Klein, Ass.-Prof. PD Dr., Medical University of Vienna
Other Study IDs: MAS 1120/2013
Record Dates: First submitted 2013-12-22; First posted 2013-12-30 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Atelectasis
Keywords: atelectasis; SPO2 - oscillations
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: None Retained — Spo2 Ventilation
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Even though experimental lung injury in animal experiments is the best analogy for the changes in the patients, it has to be considered that kinetics may vary between species. An important question to answer is how common PaO2-oscillations occur in patients and how injurious they might be. A limitation to the detection of PaO2-oscillations is a sensing device that detects the oscillations at very high temporal resolution. In previous studies a fiberoptic probe was used, which was measuring PaO2 based on oxygen-sensitive fluorescence quenching with a time resolution up to 10 Hz (8, 13, 14). This method is not feasible in patients. Previous studies have shown that PaO2-oscillations are translated into the peripheral hemoglobin oxygen saturation (SpO2). Given a technology that has a time resolution that is high enough (i.e. >1 Hz), measurement of SpO2-oscillations would be a valid approach to detecting and quantifying cyclical recruitment and derecruitment in a non-invasive fashion in patients on the ICU. The Masimo Rad-8 pulse-oxymeter provides such a method. In the current study it is planned to deteted SpO2-oscillations in the post-operative patients on the ICU.

DETAILED DESCRIPTION:
As stated above cyclical recruitment and derecruitment has been shown a mechanism of VALI. It has further been demonstrated that PaO2-oscillations in the systemic circulation are transmitted to endorgans (i.e. brain, kidney and other peripheral organs). There have no studies quantifying PaO2- or SpO2-oscillations in human subjects. The rationale of this study is to measure non-invasively SpO2-oscillations throughout the respiratory cycle as PaO2 oscillations cannot easily be detected. We will analyse SpO2-oscillations in a cohort of post-operative patients. Atelectasis is a major risk factor for pulmonary complications. As it occurs in up to 90% of surgical patients this phenomenon is highly relevant. Patients with large areas of atelectatic lung tissue are prone to cyclical recruitment and derecruitment and consecutive SpO2-oscillations.

There will be two groups of patients: One with a high risk for atelectasis and one with low risk for atelectasis. The patients are stratified by the type of surgery. Upper abdominal surgery with a duration of more than 2 hours has been shown to be an independent risk factor for atelectasis. Therefore, we chose to assign patients scheduled for abdominal surgery with an anticipated duration of surgery of more than 4 hours for the high-risk group. Patients with neurosurgical procedures with more than 4 hours will be assigned to the low risk group. In each patient the SpO2-oscillations will be measured at three different respiratory rates (RR). The rationale for this is that previous studies showed that cyclical recruitment and derecruitment is dependent on the RR.

ELIGIBILITY:
Inclusion Criteria:

Interventional group:

Patients who are at high risk of developing atelectasis at the end of the operation, i.e. having had large abdominal surgery for longer than 4 hours.

Control group:

Patients who are at low risk of developing atelectasis at the end of the operation, i.e. having had neurosurgical treatment without opening the abdomen

Exclusion Criteria:

Interventional + control group:

Age < 18yr, alcohol or drug abuse, pregnancy, participation in another study, skin lesions on the fingers, allergy to patches or other severe allergies, patients who cannot give their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients in 2 groups
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of SpO2-oscillations caused by cyclic recruitment and derecruitment of atelectasis. | 20 min
  Desaturation of SpO2

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Ulrich Klein, PD MD, Principal Investigator — MUW/AKH
Locations (1):
- MUW/AKH, Vienna, Austria